CLINICAL TRIAL: NCT01838291
Title: Active Drug Surveillance Program of Ferriprox Use
Status: Completed | Type: Observational
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Other Study IDs: LA35-PM
Record Dates: First submitted 2013-04-15; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Transfusional Iron Overload
Keywords: Ferriprox; Deferiprone; DFP; L1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients on Ferriprox therapy <1 month

SUMMARY:
Observational, open label, prospective, multi-center, post-marketing drug surveillance program.

DETAILED DESCRIPTION:
A post-marketing, drug surveillance program evaluating the use, monitoring, benefits and adverse effects of Ferriprox under clinical conditions in newly treated patients.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients who started Ferriprox therapy less than one month or are to initiate Ferriprox therapy at the time of enrolment into the program.

Main Exclusion Criteria:

* Patients treated with Ferriprox for more than one month prior to enrolment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Apporximately 300 patients who have recently started treatment with treatment with Ferriprox (less than one month prior to enrolment) or who are naive to Ferriprox treatment.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of dose of Ferriprox, and if applicable concurrent chelator(s) in newly treated patients. | Baseline to 12 Months
  Evaluation of dose of Ferriprox includes the frequency of administration of chelator(s).
Evaluation of regimen of Ferriprox administration, and if applicable concurrent chelator(s) in newly treated patients. | Baseline to 12 Months
  Evaluation of how Ferriprox is prescribed/received by the patient: as monotherapy, simultaneous with deferoxamine, alternate with deferoxamine, simultaneous with deferasirox, alternate with deferasirox.

SECONDARY OUTCOMES:
Assessment of the beneficial effects of Ferriprox based on the characterization of its use in clinical practice. | Baseline to 12 Months
  Beneficial effects of Ferriprox will be assessed based on the changes in: serum ferritin and cardiac iron concentration as assessed by MRI T2*.
Assessment of the adverse effects of Ferriprox based on the characterization of its use in clinical practice. | Baseline to 12 Months
  Adverse effects of Ferriprox will be assessed based on: frequency of absolute neutrophil count (ANC) monitoring, occurrence of neutropenia or agranulocytosis and occurrence of other adverse events (AEs) or adverse drug reactions (ADRs).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Tricta, MD, Study Chair — ApoPharma
Locations (14):
- Thalassemia Center of North Cyprus Turkish Republic (KKTC), Nicosia, Cyprus
- Egypt (7):
  - Hematology Unit, Mansoura University Children Hospital, Al Mansurah
  - Hematology Unit, El-Shatby Children Hospital, Alexandria University, Alexandria
  - Hematology Unit, Assiut University Hospital, Asyut
  - Ain Shams University, Cairo
  - Tanta University Hospital, Tanta
  - Hematology/Oncology Unit ; Zagazig University Children Hospital, Zagazig
  - Zagazig University; Thalassemia Association, Zagazig
- Department of Child Health, College of Medicine and Health Sciences, Sultan Qaboos University Hospital, Muscat, Oman
- Saudi Arabia (2):
  - King Abdulaziz University Hospital (KAAUH), Jeddah
  - Maternity and Children's Hospital, Maddinah
- Turkey (Türkiye) (3):
  - Çukurova Üniversitesi Tip Fakültesi, Çocuk Hematolojie Bilim Dali, Adana
  - Akdeniz Üniversitesi Hastanesi, Çocuk Sağliği, Hematolojie Kliniği, Antalya
  - Ïstanbul Üniversitesi Tip. Fak. Hastanesi, Çocuk Sağliği, Hematolojie Kliniği, Istanbul